CLINICAL TRIAL: NCT00246857
Title: Screening Protocol for Genetic Diseases of Lymphocyte Homeostasis and Programmed Cell Death
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060015; 06-I-0015
Record Dates: First submitted 2005-10-29; First posted 2005-10-31 (Estimated); Last update posted 2026-01-21 (Actual); Status verified 2026-01-16

CONDITIONS: Primary Immune Deficiency
Keywords: Apoptosis; T-cell; Autoimmunity; Lymphoproliferation; B-Cell; Inherited Lymphhocyte Homeostasis; Genetic Disease
MeSH Terms: conditions — Primary Immunodeficiency Diseases; Autoimmune Diseases; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients referred by physician with a suspected inherited immune deficiency: patients referred by physician with a suspected inherited immune deficiency

SUMMARY:
This study will determine the biochemical and genetic causes of inherited immune diseases affecting lymphocyte homeostasis. Lymphocytes are a type of white blood cell that fights infections. Normally, the body keeps a precise balance in which lymphocyte growth is matched by lymphocyte death. People with constantly enlarged lymph nodes or spleen, along with autoimmune disease, immunodeficiency, lymphoma, or other immune problems affecting lymphocytes may have an abnormality of the immune system in the cell growth and cell death processes that regulate lymphocyte homeostasis.

Patients who have, or are suspected of having, an inherited lymphocyte homeostasis or programmed cell death susceptibility syndrome may be eligible for this study. Relatives of patients are also included.

Participants' (patients and relatives) medical records are reviewed and blood samples are drawn for studies to identify genes involved in immune disorders. Tissues that have been removed from patients for medical reasons, such as biopsied tissues, may be examined for tissue and DNA studies. Relatives are studied to determine if some of them may have a very mild form of lymphocyte homeostasis disorder.

Patients who have an immune problem that the researchers wish to study further will be invited to donate additional blood samples at irregular intervals (at least once a year) and to provide an update of their medical records at the same time.

...

DETAILED DESCRIPTION:
This protocol is designed to screen patients with suspected or identified genetic diseases of immune cell homeostasis, reflecting abnormalities in programmed cell death, survival, development, activation, and/or proliferation. Patients determined by clinical history and initial outside evaluation by their referring physician to be of interest will be consented and enrolled into this study. Blood and other biological specimens from patients or their family members will be obtained for research studies related to understanding the genetic and biochemical bases of these diseases. Outside medical records will be obtained for chart review to correlate clinical history to research laboratory testing results. Results will be relayed to the referring physicians and, where applicable, patients may be referred to other relevant research studies at the NIH.

The study will enroll up to 5000 patients and family members over the next 20 years.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients known to have or suspected of having an inherited immune cell homeostasis, programmed cell death susceptibility syndrome, lymphocyte developmental block, or defective immune cell effector functions will be eligible for enrollment. We will enroll

patients with suspected disease if the investigator agrees that there is a high index of suspicion. Blood relatives of enrolled patients will be eligible for enrollment. There will be no limit as to age, sex, race, or disability.

EXCLUSION CRITERIA:

Severely debilitated health status or poor venous access may preclude obtaining adequate specimens for analysis. The minimum weight for infants on this protocol is 3 kg because of the limits of maximal acceptable blood draw volumes and minimum requirement for core laboratory tests would exceed the acceptable volume.

Ages: 1 Month to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients referred by physician with a suspected inherited immune deficiency and their unaffected relatives.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2007-02-12 (Actual)

PRIMARY OUTCOMES:
determination of underlying susceptibility trait(s) and elucidation of its mechanism of action | 2030
  Goal of this study is to determine the molecular, genetic, biochemical basis for an immune problem.

CONTACTS AND LOCATIONS:
Overall Officials: Helen C Su, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (7):
- United States (2):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - University of Michigan, Ann Arbor, Michigan
- Turkey (Türkiye) (5):
  - Ankara Medical University, Ankara
  - Gazi University, Ankara
  - Hacettepe University, Ankara
  - Marmara University, Istanbul
  - Necemttin Erbakan University, Konya

IPD SHARING:
Plan to Share IPD: No
If an individual requests to have their raw sequencing data, we have asked the IRB for permission. This has happened in one case. @@@@@@@@@@@@In another case during this reporting period, a subject asked us to share raw sequencing data with an academic center for analysis. This required a DTA which was recently completed.@@@@@@@@@@@@Sequencing is done under research conditions and is not shared with a subject unless it is verified with a repeat independent sample and CLIA certified.

REFERENCES:
- [Background] Lo B, Zhang K, Lu W, Zheng L, Zhang Q, Kanellopoulou C, Zhang Y, Liu Z, Fritz JM, Marsh R, Husami A, Kissell D, Nortman S, Chaturvedi V, Haines H, Young LR, Mo J, Filipovich AH, Bleesing JJ, Mustillo P, Stephens M, Rueda CM, Chougnet CA, Hoebe K, McElwee J, Hughes JD, Karakoc-Aydiner E, Matthews HF, Price S, Su HC, Rao VK, Lenardo MJ, Jordan MB. AUTOIMMUNE DISEASE. Patients with LRBA deficiency show CTLA4 loss and immune dysregulation responsive to abatacept therapy. Science. 2015 Jul 24;349(6246):436-40. doi: 10.1126/science.aaa1663. PMID 26206937
- [Background] Afzali B, Gronholm J, Vandrovcova J, O'Brien C, Sun HW, Vanderleyden I, Davis FP, Khoder A, Zhang Y, Hegazy AN, Villarino AV, Palmer IW, Kaufman J, Watts NR, Kazemian M, Kamenyeva O, Keith J, Sayed A, Kasperaviciute D, Mueller M, Hughes JD, Fuss IJ, Sadiyah MF, Montgomery-Recht K, McElwee J, Restifo NP, Strober W, Linterman MA, Wingfield PT, Uhlig HH, Roychoudhuri R, Aitman TJ, Kelleher P, Lenardo MJ, O'Shea JJ, Cooper N, Laurence ADJ. BACH2 immunodeficiency illustrates an association between super-enhancers and haploinsufficiency. Nat Immunol. 2017 Jul;18(7):813-823. doi: 10.1038/ni.3753. Epub 2017 May 22. PMID 28530713
- [Background] Ozen A, Comrie WA, Ardy RC, Dominguez Conde C, Dalgic B, Beser OF, Morawski AR, Karakoc-Aydiner E, Tutar E, Baris S, Ozcay F, Serwas NK, Zhang Y, Matthews HF, Pittaluga S, Folio LR, Unlusoy Aksu A, McElwee JJ, Krolo A, Kiykim A, Baris Z, Gulsan M, Ogulur I, Snapper SB, Houwen RHJ, Leavis HL, Ertem D, Kain R, Sari S, Erkan T, Su HC, Boztug K, Lenardo MJ. CD55 Deficiency, Early-Onset Protein-Losing Enteropathy, and Thrombosis. N Engl J Med. 2017 Jul 6;377(1):52-61. doi: 10.1056/NEJMoa1615887. Epub 2017 Jun 28. PMID 28657829
- [Derived] Comrie WA, Faruqi AJ, Price S, Zhang Y, Rao VK, Su HC, Lenardo MJ. RELA haploinsufficiency in CD4 lymphoproliferative disease with autoimmune cytopenias. J Allergy Clin Immunol. 2018 Apr;141(4):1507-1510.e8. doi: 10.1016/j.jaci.2017.11.036. Epub 2018 Jan 2. No abstract available. PMID 29305315
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2006-I-0015.html